CLINICAL TRIAL: NCT02173756
Title: Evaluation of Oral Morphine Gel in Oral Mucositis Induced by Chemotherapy in Children and Young Adults
Acronym: MorphinOgel
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Numerous premature study discontinuations due to adverse events
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5092
Record Dates: First submitted 2014-06-14; First posted 2014-06-25 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2014-06

CONDITIONS: Cancer
Keywords: chemotherapy; mucositis; systemic opioids; morphine
MeSH Terms: conditions — Neoplasms; Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral morphine gel (Experimental): 1 mg / ml of Morphine hydrochloride, presented in a 5 mL sterile syringe (single dose). Gel will be applied 8 times per day and for the duration of the mucositis (between 8 to 21 days).
  Interventions: Drug: morphine gel
- placebo gel (Placebo Comparator): 1 mg / ml of Placebo gel that is presented in a 5 mL sterile syringe (single dose). Gel will be applied 8 times per day and for the duration of the mucositis (between 8 to 21 days).
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: morphine gel — 1 mg / ml ofmorphine hydrochloride, presented in a 5 mL sterile syringe (single dose), raspberry aroma, 30% glucose
  Other Names: Morphine hydrochloride,
  Arms: oral morphine gel
Drug: placebo gel — Sterile placebo gel with raspberry aroma, 30% glucose presented in 5 mL syringe (single dose) of the same appearance and the same packaging as morphine gel to maintain the blind
  Other Names: sterile Placebo gel
  Arms: placebo gel

SUMMARY:
Chemotherapy kills tumor cells but can also damage healthy cells and cause significant digestive disorders such as ulcers of the mouth, called mucositis. Mucositis are transient but their intensity may require special measures. Mucositis are painful and morphine gel or intravenous morphine is used to relieve pain.

However, the pain of oral mucositis induced by chemotherapy is not completely relieved by morphine administered intravenously.

As part of the study, the investigators want to evaluate an oral gel containing a small amount of morphine so that it acts directly on the mucositis. The investigators believe that the direct action of morphine on mucositis may be more effective on pain.

DETAILED DESCRIPTION:
The objective of the study is to compare the analgesic efficacy of topical morphine gel versus placebo gel in the pediatric oncohaematology oral mucositis induced by chemotherapy in children treated with systemic opioids.

To confirm these results, we propose to conduct a randomized double-blinded study designed to compare the analgesic efficacy of morphine oral topical gel versus placebo gel in children over 5 years with mucositis induced by chemotherapy and treated with systemic opioids. This analgesic effect should reduce persistent pain to maintain oral feeding and thus delay the implementation of parenteral nutrition, and hence reduce the dose of systemic morphine and also reduce the adverse effects of opioids

ELIGIBILITY:
Inclusion Criteria:

* Children older than 5 years or adults over 18 and up to 25 years with a chemotherapy
* greater than or equal to grade 2 mucositis that has lasted for 24 hours and treated with systemic opioid

Exclusion Criteria:

* Patients in emergency ward -Patients having difficulties in understanding the study -
* Patients who have already been treated with oral morphine gel

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
change in pain of mucositis before and after meal | Daily assessment through out the mucositis
  Pain is assessed before gel application and 30 minutes after application (i e 8 times per day and for the duration of the mucositis between 8 to 21 days). The gel is administered 4 times daily 30 minutes before each meal. Response to treatment is defined as a greater than or equal to 30% decrease in pain level between before and after application of the gel.

SECONDARY OUTCOMES:
Evaluation of the local tolerance and other topical treatment taken throughout the mucositis | daily, 8-21 days throughout the mucositis
  Evaluation of the local tolerance ( taste, burns) with a questionnaire
Evaluation of the local tolerance and other topical treatment taken throughout the mucositis | daily, 8-21 days throughout the mucositis
  Assessment of the quantity of morphine in mg/ day (reported in mg morphine), the nature and amount of all systemic analgesics
Evaluation of the local tolerance and other topical treatment taken throughout the mucositis | daily, 8-21 days throughout the mucositis
  Daily grading of mucositis by the doctor
Evaluation of the local tolerance and other topical treatment taken throughout the mucositis | daily, 8-21 days throughout the mucositis
  Daily evaluation of other topical treatments administered (mouthwashes: time frames when administered, doses, nature)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'oncohématologie pédiatrique, Hôpital de Hautepierre, Strasbourg, Alsace, France